CLINICAL TRIAL: NCT01125215
Title: Study of Topical Preparation of Capsaicin Nanoparticle in Patient With Painful Diabetic Neuropathy
Brief Title: Capsaicin Nanoparticle in Patient With Painful Diabetic Neuropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Pongsatorn Meesawatsom, Mr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUPYPM-01
Record Dates: First submitted 2010-05-15; First posted 2010-05-18 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Painful diabetic neuropathy; Capsaicin; Nanoparticle; Quantitative Sensory Testing
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matched gel base of capsaicin nanoparticle
  Interventions: Drug: Placebo
- Capsaicin (Experimental): 0.075% capsaicin nanoparticle gel
  Interventions: Drug: 0.75% capsaicin nanoparticle cream

INTERVENTIONS:
Drug: 0.75% capsaicin nanoparticle cream — 0.75% capsaicin nanoparticle cream apply to area with neuropathic pain twice daily for 12 weeks
  Arms: Capsaicin
Drug: Placebo — Identical cream base of nanoparticle apply to area with neuropathic pain twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The objectives of this study are to determine efficacy and safety of 0.75% topical capsaicin nanoparticle preparation versus placebo in patient with painful diabetic neuropathy.

DETAILED DESCRIPTION:
Painful diabetic neuropathy is the most common cause of neuropathic pain. 0.075% topical capsaicin has been used to treat the pain. Because of high concentration, conventional capsaicin topical preparation causing burning sensation and required several time of applications per day.

The nanoparticle of capsaicin topical preparation was developed with expectation of remaining efficacy, minimizing burning sensation and improving convenience of use.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 Diabetes mellitus
* Peripheral neuropathy
* Stabilized on pain medication for at least one month
* No previous invasive intervention for pain relief

Exclusion Criteria:

* Local wound or any skin abnormality in the applicable area
* Allergic to capsaicin
* Refuse to participate or give consent
* Has other significant disease or receive medication that may worsen neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief from pain score reduction, using visual analog scale (VAS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chuthamanee Suthisisang, PhD., Study Director — Faculty of Pharmacy,Mahidol University
Locations (2):
- Thailand (2):
  - Ramathibodi Hospital, Bangkok, Bangkok
  - Thammasat University Hospital, Pathum Thani, Changwat Pathum Thani